CLINICAL TRIAL: NCT01298960
Title: Phase II Randomized Study of Cotreatment With Growth Hormone in a Long GnRH Agonist Protocol in Women With Previous Poor Ovarian Response
Brief Title: Growth Hormone (GH) in in Vitro Fertilization (IVF) Poor-responder Patients
Acronym: FUNDEX001
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Principal Investigator, Ignacio Rodriguez MSc, BSC, Fundacion Dexeus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUNDEX001; 2010-022151-32 (EudraCT Number)
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Complications; Artificial Fertilization, Introduction of Embryo in Embryo Transfer
Keywords: Poor Ovarian response in IVF; Metaphase II oocytes; Pregnancy Rate; Growth Hormone
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rGH Group (Experimental)
  Interventions: Drug: Somatropin
- Non rGH group (No Intervention)

INTERVENTIONS:
Drug: Somatropin — 0.1 IU/Kg/day from day one of stimulation until rHCG triggering
  Arms: rGH Group

SUMMARY:
Experimental study to evaluate if rGH addition to a standard controlled ovarian stimulation treatment improves ovarian response in women with previous poor ovarian response.

ELIGIBILITY:
Inclusion Criteria:

* Women who desire pregnancy with regular spontaneous menstrual cycles of 25-30 days length.
* Infertility requiring IVF with or without ICSI.
* Antecedent of a failed previous IVF cycle with a GnRH long agonist protocol in which at least 3000 IU of FSH were used (cancellation due to poor ovarian response - < 4 mature follicles - or less than 5 oocytes retrieved)and antral follicle count < 5.
* Partner sperm.
* Presence of both ovaries and normal uterine cavity.
* PAP smear within normality in previous 3 years.
* Negative pregnancy test (serum or urine) before rFSH administration.
* Willingness of adhesion to protocol during the whole study period.
* Signed informed consent given.

Exclusion Criteria:

* HIV, HCV, HBV positive serologies in women or partner.
* Important systemic diseases that could interfere with gonadotrophin treatment (ovarian and hypothalamic tumors...).
* BMI > 32 kg/m2 or antecedent of diabetes mellitus.
* Gonadotrophin treatment within the previous 30 days.
* Availability of frozen embryos of previous IVF cycles .
* Abnormal uterine bleeding.
* Previous treatment with LH or LH effect drugs.
* Polycystic ovaries, increased size ovaries or presence of ovarian cysts of unknown ethiology.
* Contraindication for pregnancy.
* Allergies to gonadotrophins or somatotropin.
* History of drug or alcohol abuse in the previous 5 years.
* Previous enrollment in this study or simultaneous participation in another study with drugs.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Number of metaphase II oocytes retrieved | 3 months after having finished recruitment

SECONDARY OUTCOMES:
Pregnancy rate | 9 months after ovum pick-up
Adverse events due to rGH | 3 months after having finished recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Pedro N Barri, PhD, MD, Study Chair — Department of Obstetrics, Gyneacology and Reproductive Medicine, Institut Universitari Dexeus; Buenaventura Coroleu, PhD. MD, Principal Investigator — Departament of Obstetrics, Gyneacology and Reproductive Medine, Institut Universitari Dexeus; Marta Devesa, MD, Principal Investigator — Department of Obstetrics, Gyneacology and Reproductive Medicine, Institut Universitari Dexeus; Francisca Martinez, PhD. MD, Principal Investigator — Department of Obstetrics, Gyneacology and Reproductive Medicine, Institut Universitari Dexeus
Locations (1):
- Departamento de Obstetricia Ginecologia y Reproducción. Institut Universitari Dexeus, Barcelona, Spain

REFERENCES:
- [Background] Harper K, Proctor M, Hughes E. Growth hormone for in vitro fertilization. Cochrane Database Syst Rev. 2003;(3):CD000099. doi: 10.1002/14651858.CD000099. PMID 12917883
- [Background] Kolibianakis EM, Venetis CA, Diedrich K, Tarlatzis BC, Griesinger G. Addition of growth hormone to gonadotrophins in ovarian stimulation of poor responders treated by in-vitro fertilization: a systematic review and meta-analysis. Hum Reprod Update. 2009 Nov-Dec;15(6):613-22. doi: 10.1093/humupd/dmp026. Epub 2009 Jun 26. PMID 19561136
- See also: Related Info — http://www.dexeus.com